CLINICAL TRIAL: NCT03997032
Title: A Pilot Study to Assess the Effect of a 3-month Folate Supplementation on Systemic Homocysteine Plasma Concentration and Ocular Blood Flow in Patients With Diabetes
Brief Title: A Study to Assess the Effect of a 3-month Folate Supplementation on Systemic Homocysteine Plasma Concentration and Ocular Blood Flow in Patients With Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Collaborators: Aprofol AG (Unknown)
Responsible Party: Principal Investigator, Gerhard Garhofer, Principal Investigator, Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 23022017
Record Dates: First submitted 2019-06-19; First posted 2019-06-25 (Actual); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — Ocufolin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with Diabetes (Experimental): Patients with Type 1 or Type 2 Diabetes
  Interventions: Dietary Supplement: Ocufolin

INTERVENTIONS:
Dietary Supplement: Ocufolin — Ocufolin, Aprofol AG, Switzerland Dose: 1 capsule per day

SUMMARY:
There is evidence that a folate deficiency - and as the biological consequence of the latter - higher homocysteine plasma levels are associated with an increased risk of vascular associated diseases. For the eye, it has been shown that higher intake of folate reduces the risk of vascular related diseases such as age related macular degeneration. Further studies suggest that decreased serum levels of folate and vitamin B12 may be an independent risk factor for diabetic retinopathy. The reason for the association of low folate levels and the increased risk for vascular-associated ocular diseases is not entirely clear but may be at least partially related to an impairment of local blood flow regulation in these patients.

Whether supplementation with folate may improve vascular regulation has not yet been sufficiently investigated. However, given that the potential effect size of a folate substitution on blood flow and systemic blood parameters is unclear, a proper statistical design for a large, controlled, randomized study is difficult. Thus, the present pilot study should (1) provide information about the homocysteine lowering potential of the formulation under study and (2) identify potential vascular related outcome parameters for further, larger, placebo-controlled studies and provide sufficient data to allow for a proper statistical planning for such a study.

Consequently, the current study seeks to investigate the effect of a 3-month supplementation with folate on systemic homocysteine plasma levels. Further, ocular blood flow and endothelial function in the ocular microcirculation will be assessed. For this purpose, a group of 25 patients with diabetes mellitus will be included in the study. Outcome parameters will be assessed at baseline and after a 3-month supplementation with folate.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Diabetes mellitus type 1 or 2
* No or mild non-proliferative diabetic retinopathy
* Normal findings in the medical history except diabetes unless the investigator considers an abnormality to be clinically irrelevant
* Normal ophthalmic findings except mild non-proliferative retinopathy
* Ametropy ≤ 6 diopters

Exclusion Criteria:

* Participation in a clinical trial in the 3 weeks preceding the screening visit
* Symptoms of a clinically relevant illness in the 3 weeks before the first study day
* Presence or history of a severe medical condition relevant to the study, except diabetes, as judged by the clinical investigator
* Intake of dietary supplements containing folate within the three months before the screening visit
* Untreated or uncontrolled arterial hypertension (defined as either systolic blood pressure >150 mmHg or diastolic blood pressure >95 mmHg)
* Blood donation during the previous three weeks
* Moderate to severe non-proliferative or proliferative diabetic retinopathy
* Previous laser photocoagulation treatment
* History or family history of epilepsy
* Presence of any abnormalities preventing reliable measurements in the study eye as judged by the investigator
* Best corrected visual acuity < 0.8 Snellen
* Ametropy > 6 Dpt
* Pregnancy, planned pregnancy or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-07-31 (Actual); Primary Completion 2018-03-12 (Actual); Study Completion 2018-07-17 (Actual)

PRIMARY OUTCOMES:
Plasma homocysteine level | Change from Baseline plasma homocysteine level at 3 months
  Laboratory analysis for plasma homocysteine level in µmol/L

SECONDARY OUTCOMES:
Retinal blood flow | Change from Baseline retinal blood flow at 3 months
  Retinal blood flow will be assessed using Fourier domain optical coherence tomography, providing values in µl/min
Retinal vessel diameters | Change from Baseline retinal vessel diameters at 3 months

OTHER OUTCOMES:
Intraocular pressure | Change from Baseline intraocular pressure at 3 months
  Intraocular pressure will be assessed using Goldmann Applanation Tonometry, values will be provided in mmHg

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Clinical Pharmacology, Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Schmidl D, Howorka K, Szegedi S, Stjepanek K, Puchner S, Bata A, Scheschy U, Aschinger G, Werkmeister RM, Schmetterer L, Garhofer G. A pilot study to assess the effect of a three-month vitamin supplementation containing L-methylfolate on systemic homocysteine plasma concentrations and retinal blood flow in patients with diabetes. Mol Vis. 2020 Apr 24;26:326-333. eCollection 2020. PMID 32355442